CLINICAL TRIAL: NCT02153112
Title: A Phase II, Randomized, Double-Blind, Dosage, Safety and Immunogenicity Trial of Intramuscular Norovirus GI.1/GII.4 Bivalent Virus-Like Particle Vaccine Combined With Aluminum Hydroxide Adjuvant in Children, Toddlers, and Infants
Brief Title: Safety and Immunogenicity of Norovirus GI.1/GII.4 Bivalent Virus-Like Particle (VLP) Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NOR-202; 2014-000778-20 (EudraCT Number); U1111-1154-9733 (Other: World Health Organization)
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-12

CONDITIONS: Norovirus
Keywords: Drug therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1, Group 1: 1 Dose (Experimental): Children 4 to <9 years of age received one dose of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent virus-like particle (VLP) vaccine, intramuscularly (IM) and 500 µg aluminum hydroxide on Day 1, followed by placebo matching norovirus bivalent VLP vaccine IM on Day 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150); Drug: Placebo
- Cohort 1, Group 1: 2 Doses (Experimental): Children 4 to <9 years of age received 2 doses of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide IM on Days 1 and 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150)
- Cohort 1, Group 2: 1 Dose (Experimental): Children 1 to <4 years of age received one dose of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Day 1, followed by placebo-matching norovirus bivalent VLP vaccine, IM on Day 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150); Drug: Placebo
- Cohort 1, Group 2: 2 Doses (Experimental): Children 1 to <4 years of age received 2 doses of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1 and 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150)
- Cohort 1, Group 2a: 1 Dose (Experimental): Children 1 to <4 years of age received one dose of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Day 1, followed by placebo matching norovirus bivalent VLP vaccine, IM on Day 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150); Drug: Placebo
- Cohort 1, Group 2a: 2 Doses (Experimental): Children 1 to <4 years of age received 2 doses of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1 and 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150)
- Cohort 1, Group 3: 1 Dose (Experimental): Toddlers 6 months to <1 year of age received one dose of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Day 1, followed by placebo matching norovirus bivalent VLP vaccine, IM on Day 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150); Drug: Placebo
- Cohort 1, Group 3: 2 Doses (Experimental): Toddlers 6 months to <1 year of age will receive 2 doses either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1 and 29.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150)
- Cohort 2, Group 4: 2 Doses (Experimental): Infants 6 weeks to <6 months of age received 2 doses of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) formulations of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1 and 56, followed by placebo-matching norovirus bivalent VLP vaccine, IM on Day 112.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150); Drug: Placebo
- Cohort 2, Group 4: 3 Doses (Experimental): Infants 6 weeks to <6 months of age received 3 doses of either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1, 56 and 112.
  Interventions: Biological: GI.1/GII.4 (15/15); Biological: GI.1/GII.4 (15/50); Biological: GI.1/GII.4 (50/50); Biological: GI.1/GII.4 (50/150)

INTERVENTIONS:
Biological: GI.1/GII.4 (15/15) — Norovirus GI.1/GII.4 (15 μg/15 μg) bivalent VLP vaccine combined with 500 μg aluminum hydroxide for IM injection
Biological: GI.1/GII.4 (15/50) — Norovirus GI.1/GII.4 (15 μg/50 μg) bivalent VLP vaccine combined with 500 μg aluminum hydroxide for IM injection
Biological: GI.1/GII.4 (50/50) — Norovirus GI.1/GII.4 (50 μg/50 μg) bivalent VLP vaccine combined with 500 μg aluminum hydroxide for IM injection
Biological: GI.1/GII.4 (50/150) — Norovirus GI.1/GII.4 (50 μg/150 μg) bivalent VLP vaccine combined with 500 μg aluminum hydroxide for IM injection
Drug: Placebo — Placebo saline solution
  Arms: Cohort 1, Group 1: 1 Dose; Cohort 1, Group 2: 1 Dose; Cohort 1, Group 2a: 1 Dose; Cohort 1, Group 3: 1 Dose; Cohort 2, Group 4: 2 Doses

SUMMARY:
The purpose of this study is to select the optimal formulation of the norovirus vaccine from different concentrations of virus-like particles (VLP) combined with aluminum hydroxide for further development in children.

DETAILED DESCRIPTION:
The vaccine being tested in this study is called norovirus GI.1/GII.4 bivalent virus-like particle (VLP) vaccine with aluminum hydroxide. The norovirus vaccine is being tested to assess different formulations of the vaccine that will then be further developed. This study will look at the number of antibodies to norovirus formed in children, toddlers and infants who are administered different formulations of the norovirus vaccine.

The study enrolled 840 patients. Participants will be randomly assigned (by chance) to one of ten treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

All participants in Cohort 1 will be vaccinated on Day 1 and Day 29 of the study, and all participants in Cohort 2 will be vaccinated on Day 1, Day 56, and Day 112. All treatment groups in Cohort 1 will receive either one dose of the norovirus vaccine, or two doses. One treatment group in Cohort 2 will receive 2 doses of the norovirus vaccine, and the other group will receive 3. In order to keep the treatment undisclosed to the participant and the doctor in Cohort 1, those randomized to the one-dose groups will receive the norovirus vaccine on Day 1, followed by a dose of placebo vaccine on Day 29. In order to keep the treatment arms undisclosed to the participant and the doctor in Cohort 2, those randomized to the two-dose groups will receive the norovirus vaccine on Day 1 and Day 56, followed by a dose of placebo vaccine on Day 112. Placebo vaccine is saline solution. Participants will be asked to record any symptoms that may be related to the vaccine or the injection site in a diary card for 7 days after each vaccination.

This multi-center trial will be conducted in Finland, Panama, and Colombia. The overall time to participate in this study is up to 210 days for participants in Cohort 1 and up to 293 Days for participants in Cohort 2. Participants in Cohort 1 will make 6 visits to the clinic, and participants in Cohort 2 will make 10 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged between 6 weeks and less than 9 years at the time of enrollment.
2. Are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and clinical judgment of the investigator.
3. Participants legally authorized representative (LAR) signs and dates a written, informed consent form (ICF) and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements. An assent will also be obtained according to age-appropriate country-specific regulations.
4. Participants who can comply with trial procedures and are available for the duration of the trial.

Exclusion Criteria:

1. Participants with a clinically significant active infection (as assessed by the investigator) or body temperature 38.0°C (100.4°F) or higher within 3 days of the intended date of vaccination.
2. Have received antipyretic/analgesic medications within 24 hours prior to the intended vaccine administration.
3. Known hypersensitivity or allergy to investigational vaccine (including excipients of the investigational vaccines).
4. Participants with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the ability to participate in the trial.
5. Has a history of any progressive or severe neurologic disorder, seizure disorder, or neuroinflammatory disease (eg, Guillain-Barré syndrome).
6. Known or suspected impairment/alteration of immune function, including the following:

   1. Children <18 months of age with history of repeated episodes of acute otitis media (AOM) in the first 6 months of life (AOM defined as a bulging tympanic membrane) and not to be confused with otitis media with effusion (OME).
   2. Chronic use of oral steroids (equivalent to 20 mg/day prednisone for ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1 (use of inhaled, intranasal, or topical corticosteroids is allowed).
   3. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day for ≥2 weeks) within 60 days prior to Day 1.
   4. Receipt of immunostimulants within 60 days prior to Day 1.
   5. Receipt of parenteral, epidural, or intra-articular immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Day 1 or planned during the full length of the trial.
   6. Receipt of immunosuppressive therapy within 6 months prior to Day 1.
   7. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   8. Chronic Hepatitis B or C infection.
   9. Heritable immunodeficiency.
7. Abnormalities of splenic or thymic function.
8. Has a known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
9. Has any serious chronic or progressive disease according to judgment of the investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal, or hepatic disease).
10. Is participating in any clinical trial with another investigational product 30 days prior to first trial visit or intent to participate in another clinical trial at any time during the conduct of this trial.
11. Has received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial.
12. Are first degree relatives of individuals involved in trial conduct.
13. Has a history of autoimmune disease.

Ages: 6 Weeks to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2015-06-23 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (12):
- Centro de Estudios em Infectologia Pediatrica SAS, Cali, San Fernando, Colombia
- Finland (9):
  - Espoon Rokotetutkimusklinikka, Espoo
  - Etela-Helsingin Rokotetutkimusklinikka, Helsinki
  - Ita-Helsingin Rokotetutkimusklinikka, Helsinki
  - Jarvenpaan Rokotetutkimusklinikka, Jarvenpaan
  - Oulun Rokotetutkimusklinikka, Oulu
  - Porin Rokotetutkimusklinikka, Pori
  - Seinajoen Rokotetutkimusklinikka, Seinäjoki
  - Tampere Vaccine Research Clinic, Tampere
  - Turun Rokotetutkimusklinikka, Turku
- Panama (2):
  - CEVAXIN Plaza Carolina - Ciudad de Panama, Panama City
  - CEVAXIN, Panama City

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Lopez P, Lopez-Medina E, Saez-Llorens X, deAntonio R, Masuda T, Mendelman PM, Sherwood J, Baehner F, Borkowski A. Immunogenicity and tolerability of a bivalent virus-like particle norovirus vaccine candidate in children from 6 months up to 4 years of age: A phase 2 randomized, double-blind trial. Hum Vaccin Immunother. 2023 Dec 31;19(1):2204787. doi: 10.1080/21645515.2023.2204787. Epub 2023 May 4. PMID 37140558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 12 investigative sites in Finland, Panama, and Colombia from 23 June 2015 to 20 June 2018.
Pre-assignment Details: Healthy volunteers (children, toddlers and infants) were enrolled to receive either one, two or three doses of 4 formulation of norovirus GI.1/GII4 bivalent virus like particle (VLP) vaccine.
Groups:
- Cohort 1, Group 3: 2 Doses: Toddlers 6 months to <1 year of age received 2 doses either of the 4 formulations (15 µg of GI.1 norovirus VLP and 15 µg GII.4/GI.1/GII.4 (15 μg/50 μg)/GI.1/GII.4 (50 μg/50 μg) or GI.1/GII.4 (50 μg/150 μg) of the norovirus bivalent VLP vaccine and 500 µg aluminum hydroxide, IM on Days 1 and 29.
Period: Overall Study
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Started | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 180
Completed | 57 | 57 | 58 | 57 | 57 | 58 | 52 | 58 | 165 | 166
Not Completed | 4 | 2 | 3 | 2 | 3 | 2 | 8 | 2 | 15 | 14
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 2 | 1 | 1 | 7 | 2 | 13 | 12
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Per-Protocol Analysis Set (PPS) included all participants who received the planned vaccination and do not have major protocol violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses | Total
Number analyzed (Participants) | 54 | 54 | 55 | 57 | 52 | 56 | 52 | 56 | 144 | 162 | 742
Age, Continuous [Mean (Full Range); unit: years] | 5.9 [4 to 8] | 5.8 [4 to 8] | 2.1 [1 to 3] | 2.1 [1 to 3] | 1.9 [1 to 3] | 2.1 [1 to 3] | 8.3 [6 to 11] | 7.9 [6 to 11] | 3.1 [1 to 5] | 3.0 [1 to 5] | 4.22 [1 to 11]
Age, Customized [Count of Participants; unit: Participants]
  EU Registration Age Categories: Infants and Toddlers (28 days-23 months) | 0 | 0 | 17 | 19 | 15 | 14 | 52 | 56 | 144 | 162 | 479
  EU Registration Age Categories: Children (2-11 years) | 54 | 54 | 38 | 38 | 37 | 42 | 0 | 0 | 0 | 0 | 263
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 27 | 25 | 28 | 19 | 24 | 27 | 77 | 72 | 355
  Male | 22 | 30 | 28 | 32 | 24 | 37 | 28 | 29 | 67 | 90 | 387
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 24 | 26 | 29 | 52 | 56 | 52 | 56 | 144 | 162 | 627
  Not Hispanic or Latino | 28 | 30 | 28 | 27 | 0 | 0 | 0 | 0 | 0 | 0 | 113
  Not Reported | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 19 | 9 | 9 | 11 | 10 | 24 | 29 | 69 | 75 | 273
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 1 | 0 | 0 | 8 | 10 | 7 | 5 | 16 | 24 | 73
  Native Hawaiian or Other Pacific Islanders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 28 | 30 | 28 | 27 | 0 | 2 | 2 | 0 | 1 | 3 | 121
  Multiracial | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 6 | 4 | 17 | 20 | 33 | 34 | 17 | 22 | 58 | 60 | 271
Height [Mean (Full Range); unit: cm] | 117.4 [92 to 138] | 116.5 [96 to 138] | 89.9 [67 to 105] | 89.8 [73 to 104] | 89.7 [74 to 117] | 89.9 [72 to 110] | 70.6 [63 to 80] | 69.3 [64 to 75] | 60.2 [50 to 71] | 60.2 [51 to 68] | 85.35 [50 to 138]
Weight [Mean (Full Range); unit: kg] | 22.41 [13.7 to 43.2] | 22.19 [13.6 to 45.3] | 13.55 [8.0 to 19.4] | 13.39 [10.0 to 18.6] | 13.19 [8.8 to 17.5] | 13.11 [8.9 to 21.8] | 9.02 [6.0 to 14.0] | 8.85 [6.2 to 11.1] | 6.33 [3.5 to 9.5] | 6.35 [3.4 to 9.5] | 12.839 [3.4 to 45.3]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Seroresponse (Pan-Ig ELISA) in Cohort 1
Description: Seroresponse was defined as 4-fold rise or greater at Day 57 in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 57
Population: Per-protocol set included all participants who received the planned vaccination and do not have major protocol violations. Overall number of participants analyzed is the number of participants with data available at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55
percentage of participants | 77.4 [63.8 to 87.7] | 63.5 [49.0 to 76.4] | 74.5 [60.4 to 85.7] | 85.7 [73.8 to 93.6] | 53.2 [38.1 to 67.9] | 70.4 [56.4 to 82.0] | 71.4 [56.7 to 83.4] | 92.7 [82.4 to 98.0]

2. Primary Outcome: Percentage of Participants With a Seroresponse (Pan-Ig ELISA) in Cohort 2
Description: Seroresponse was defined as 4-fold rise or greater at Day 140 in serum anti-norovirus antibody titers for both GI.1 virus-Like particle (VLP) and GII.4 VLP as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 131 | 146
percentage of participants | 57.3 [48.3 to 65.9] | 84.9 [78.1 to 90.3]

3. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 1
Description: Solicited local AEs at injection site are defined as: pain, erythema, induration, and swelling that occur on the vaccination day through Day 7 after each vaccination.
Time Frame: Day 1 after either of the vaccination given on Days 1, 29, 56 or 112
Population: Safety analysis set included all participants who received at least 1 dose of vaccine (NoV GI.1/GII.4 bivalent VLP vaccine or control vaccine). Overall number of participants analyzed is the number of participants with data available at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
percentage of participants
  Any solicited local AEs | 52.5 | 66.1 | 34.4 | 45.8 | 26.7 | 30.0 | 11.7 | 13.3 | 22.2 | 30.7
  Pain | 52.5 | 66.1 | 34.4 | 35.6 | 26.7 | 25.0 | 8.3 | 13.3 | 22.2 | 28.5
  Erythema | 0 | 1.7 | 1.6 | 0 | 0 | 1.7 | 3.3 | 0 | 1.1 | 2.8
  Induration | 1.6 | 1.7 | 0 | 1.7 | 0 | 1.7 | 1.7 | 0 | 0 | 0
  Swelling | 0 | 5.1 | 0 | 0 | 0 | 1.7 | 0 | 0 | 0.6 | 0

4. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 2
Description: as for outcome 3
Time Frame: Day 1 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 178
percentage of participants
  Any solicited local AEs | 41.0 | 44.1 | 8.2 | 25.4 | 13.3 | 15.0 | 10.0 | 5.0 | 13.3 | 14.5
  Pain | 41.7 | 44.8 | 6.6 | 23.7 | 13.3 | 13.3 | 6.9 | 5.1 | 13.6 | 14.6
  Erythema | 0 | 0 | 3.3 | 5.1 | 0 | 0 | 1.7 | 0 | 0.6 | 0
  Induration | 0 | 0 | 0 | 1.7 | 0 | 1.7 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 1.7 | 0 | 1.7 | 1.7 | 0 | 0.6 | 0

5. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 3
Description: as for outcome 3
Time Frame: Day 3 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 178
percentage of participants
  Any solicited local AEs | 13.1 | 15.3 | 4.9 | 20.3 | 10.0 | 10.0 | 5.0 | 6.7 | 2.2 | 5.0
  Pain | 13.3 | 15.5 | 4.9 | 20.3 | 10.0 | 8.3 | 3.4 | 6.8 | 2.3 | 5.1
  Erythema | 0 | 0 | 1.6 | 3.4 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 1.6 | 0 | 0 | 1.7 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 1.6 | 3.4 | 0 | 1.7 | 1.7 | 0 | 0 | 0

6. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 4
Description: as for outcome 3
Time Frame: Day 4 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 178
percentage of participants
  Any solicited local AEs | 6.6 | 6.8 | 1.6 | 11.9 | 6.7 | 10.0 | 6.7 | 6.7 | 3.3 | 4.5
  Pain | 6.7 | 6.9 | 0 | 11.9 | 6.7 | 6.7 | 5.2 | 6.8 | 3.4 | 4.5
  Erythema | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 1.6 | 1.7 | 0 | 1.7 | 1.7 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 1.7 | 0 | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 5
Description: as for outcome 3
Time Frame: Day 5 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 178
percentage of participants
  Any solicited local AEs | 0 | 5.1 | 1.6 | 5.1 | 3.3 | 1.7 | 3.3 | 8.3 | 1.7 | 2.8
  Pain | 0 | 5.2 | 0 | 5.1 | 3.3 | 1.7 | 3.4 | 8.5 | 1.7 | 2.8
  Erythema | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 1.6 | 1.7 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 6
Description: as for outcome 3
Time Frame: Day 6 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 179
percentage of participants
  Any solicited local AEs | 3.3 | 3.4 | 0 | 3.4 | 1.7 | 1.7 | 1.7 | 5.0 | 1.1 | 4.5
  Pain | 3.3 | 3.4 | 0 | 3.4 | 1.7 | 1.7 | 1.7 | 5.1 | 0.6 | 4.5
  Erythema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 0 | 1.7 | 0 | 0 | 0 | 1.7 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination on Day 7
Description: as for outcome 3
Time Frame: Day 7 after either of the vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 60 | 58 | 61 | 59 | 60 | 60 | 58 | 59 | 176 | 178
percentage of participants
  Any solicited local AEs | 1.6 | 3.4 | 0 | 1.7 | 1.7 | 1.7 | 1.7 | 3.3 | 0.6 | 2.2
  Pain | 1.7 | 3.4 | 0 | 1.7 | 1.7 | 1.7 | 1.7 | 3.4 | 0.6 | 2.2
  Erythema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Induration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) (Diary-Recorded) Following Either Vaccination
Description: Systemic AEs are defined as headache, fatigue, myalgia, arthralgia, vomiting (number per day/intensity), and diarrhea (number per day/consistency) for children aged 4 to <9 years; and irritability/fussiness, drowsiness, loss of appetite, vomiting (number per day/intensity), and diarrhea (number per day/consistency) for children aged 6 weeks to <4 years on the day of vaccination and daily through Day 7 after each vaccination.
Time Frame: Days 1 through 7 after each vaccination given on Days 1, 29, 56 or 112
Population: Safety analysis set included all participants who received at least 1 dose of vaccine (NoV GI.1/GII.4 bivalent VLP vaccine or control vaccine).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
percentage of participants
  Any solicited systemic AEs | 50.8 | 61.0 | 44.3 | 54.2 | 41.7 | 43.3 | 56.7 | 50.0 | 60.0 | 59.2
  Headache | 21.7 | 25.9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 23.3 | 29.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia | 26.7 | 24.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia | 1.7 | 6.9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vomiting | 8.3 | 5.2 | 6.6 | 6.8 | 10.0 | 11.7 | 27.6 | 16.9 | 21.6 | 23.6
  Diarrhea | 6.9 | 10.7 | 13.1 | 23.7 | 18.3 | 18.3 | 31.0 | 25.4 | 31.8 | 30.9
  Irritability/Fussiness | 0 | 0 | 23.0 | 30.5 | 23.3 | 18.3 | 27.6 | 23.7 | 40.3 | 41.6
  Drowsiness | 0 | 0 | 16.4 | 22.0 | 23.3 | 21.7 | 22.4 | 20.3 | 33.5 | 33.1
  Loss of Appetite | 0 | 0 | 21.3 | 33.9 | 16.7 | 18.3 | 25.9 | 23.7 | 22.7 | 19.7

11. Primary Outcome: Body Temperature Through Day 7 Following Either Vaccination
Description: Body temperature measurement was performed using the thermometer provided by the site through Day 7 after each vaccination. The highest body temperature observed each day was recorded on the Diary Card. Body temperature is categorized as 1) Any (temperature 38°C or higher), 2) 38°C - <38.5°C, 3) 38.5°C - <39°C, 4) 39°C - <39.5°C, 5) 39.5°C - <40°C, 6) 40°C or higher. Number of participants with the particular body temperature is reported within the pre-defined categories.
Time Frame: Post-vaccination approximately 30 minutes and 6 hours later, then daily through Day 7 after each vaccination given on Days 1, 29, 56 or 112
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
participants
  Any (temperature 38°C or higher) | 2 | 6 | 7 | 5 | 6 | 8 | 8 | 11 | 26 | 23
  38°C - <38.5°C | 0 | 2 | 2 | 3 | 4 | 4 | 5 | 4 | 13 | 11
  38.5°C - <39°C | 1 | 2 | 3 | 2 | 1 | 3 | 3 | 2 | 12 | 7
  39°C - <39.5°C | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 3
  39.5°C - <40°C | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
  40°C or higher | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Percentage of Participants With at Least One Unsolicited AE Following Either Vaccination Dose
Description: Unsolicited AEs are any local or systemic AEs, as defined by this study, that are not solicited.
Time Frame: Unsolicited AEs were collected within 28 days of all vaccinations (Day 1 to 57 for Cohort 1 and Day 1 to 140 for Cohort 2)
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
percentage of participants | 55.7 | 55.9 | 67.2 | 69.5 | 55.0 | 46.7 | 73.3 | 70.0 | 77.2 | 76.0

13. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Cohort 1: Day 1 up to Day 210; Cohort 2: Day 1 up to Day 293
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
percentage of participants | 1.6 | 3.4 | 1.6 | 3.4 | 10.0 | 1.7 | 10.0 | 8.3 | 9.4 | 13.4

14. Secondary Outcome: Percentage of Participants With a Seroresponse for GI.1 Virus-Like Particle (VLP) (Pan-Ig ELISA)
Description: Seroresponse was defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-Like particle (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: Per-protocol set included all participants who received the planned vaccination and do not have major protocol violations. Here, overall number of participants analyzed is the number of participants with data available at the given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 138 | 150
percentage of participants | 88.7 [77.0 to 95.7] | 82.7 [69.7 to 91.8] | 92.2 [81.1 to 97.8] | 92.9 [82.7 to 98.0] | 78.7 [64.3 to 89.3] | 94.4 [84.6 to 98.8] | 95.9 [86.0 to 99.5] | 100.0 [93.5 to 100.0] | 94.9 [89.8 to 97.9] | 98.0 [94.3 to 99.6]

15. Secondary Outcome: Percentage of Participants With a Seroresponse for GII.4 Virus-Like Particle (VLP) (Pan-Ig ELISA)
Description: Seroresponse was defined as 4-fold rise or greater in serum anti-norovirus antibody titers for GII.4 virus-Like particle (VLP) as measured by pan immunoglobulin (Pan-Ig) enzyme-linked immunosorbent assay (ELISA).
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 134 | 150
percentage of participants | 81.1 [68.0 to 90.6] | 69.2 [54.9 to 81.3] | 76.5 [62.5 to 87.2] | 87.5 [75.9 to 94.8] | 63.8 [48.5 to 77.3] | 72.2 [58.4 to 83.5] | 75.5 [61.1 to 86.7] | 92.7 [82.4 to 98.0] | 58.2 [49.4 to 66.7] | 86.0 [79.4 to 91.1]

16. Secondary Outcome: Geometric Mean Titer (GMT) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GI.1 VLP antibody titers as measured by pan-Ig ELISA.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 144 | 162
titer | 6039.1 [4786.3 to 7619.9] | 12907.6 [10875.5 to 15319.4] | 2856.2 [2232.0 to 3654.9] | 7350.8 [6208.6 to 8703.2] | 3892.1 [2852.7 to 5310.3] | 12623.8 [10074.0 to 15818.9] | 1240.1 [948.3 to 1621.7] | 7139.1 [5863.5 to 8692.2] | 4121.1 [3688.4 to 4604.6] | 11806.3 [10537.6 to 13227.8]

17. Secondary Outcome: Geometric Mean Titer (GMT) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean titer (GMT) of anti-norovirus GII.4 VLP antibody titers as measured by pan-Ig ELISA.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 143 | 162
titer | 11057.9 [8257.3 to 14808.3] | 10228.3 [8171.2 to 12803.3] | 3293.0 [2220.5 to 4883.3] | 7955.2 [6065.9 to 10433.0] | 5950.6 [3927.2 to 9016.7] | 10896.5 [8452.0 to 14048.0] | 620.2 [383.7 to 1002.7] | 3252.1 [2403.3 to 4400.7] | 1316.2 [1103.9 to 1569.4] | 3829.8 [3311.7 to 4428.9]

18. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GI.1 VLP antibody titers as measured by pan-Ig ELISA. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 138 | 150
ratio | 19.22 [12.98 to 28.44] | 43.55 [25.21 to 75.25] | 44.11 [28.48 to 68.32] | 89.95 [56.51 to 143.18] | 13.01 [7.92 to 21.37] | 43.99 [27.71 to 69.83] | 47.45 [30.59 to 73.60] | 276.41 [206.44 to 370.09] | 34.11 [26.54 to 43.84] | 122.80 [93.93 to 160.54]

19. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (Pan-Ig ELISA)
Description: Geometric mean fold rise (GMFR) of anti-norovirus GII.4 VLP antibody titers as measured by pan-Ig ELISA. The fold rise was calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 53 | 52 | 51 | 56 | 47 | 54 | 49 | 55 | 134 | 150
ratio | 7.46 [5.63 to 9.87] | 10.00 [6.74 to 14.85] | 10.87 [7.48 to 15.77] | 19.20 [12.66 to 29.11] | 5.62 [3.83 to 8.22] | 11.93 [7.46 to 19.07] | 9.54 [5.80 to 15.71] | 55.73 [36.50 to 85.09] | 7.85 [5.86 to 10.50] | 23.55 [17.85 to 31.08]

20. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum Antibody Titers for GI.1 VLP and GII.4 VLP (HBGA)
Description: Percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for both GI.1 VLP and GII.4 VLP as measured by histoblood group antigen (HBGA) binding assay.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 48 | 47 | 44 | 49 | 43 | 47 | 30 | 41 | 129 | 144
percentage of participants | 75.0 [60.4 to 86.4] | 91.5 [79.6 to 97.6] | 50.0 [34.6 to 65.4] | 95.9 [86.0 to 99.5] | 51.2 [35.5 to 66.7] | 89.4 [76.9 to 96.5] | 36.7 [19.9 to 56.1] | 85.4 [70.8 to 94.4] | 48.1 [39.2 to 57.0] | 67.4 [59.1 to 74.9]

21. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GI.1 VLP Antibody Titers (HBGA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GI.1 virus-like particle (VLP) as measured by HBGA binding assay.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 52 | 50 | 49 | 53 | 43 | 50 | 40 | 50 | 137 | 157
percentage of participants | 94.2 [84.1 to 98.8] | 98.0 [89.4 to 99.9] | 81.6 [68.0 to 91.2] | 100.0 [93.3 to 100.0] | 74.4 [58.8 to 86.5] | 98.0 [89.4 to 99.9] | 50.0 [33.8 to 66.2] | 96.0 [86.3 to 99.5] | 92.0 [86.1 to 95.9] | 94.9 [90.2 to 97.8]

22. Secondary Outcome: Percentage of Participants With a 4-Fold Rise or Greater in Serum GII.4 VLP Antibody Titers (HBGA)
Description: The percentage of participants with a 4-fold rise or greater in serum anti-norovirus antibody titers for GII.4 virus-like particle (VLP) as measured by HBGA binding assay.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 49 | 48 | 45 | 49 | 47 | 51 | 38 | 46 | 134 | 147
percentage of participants | 81.6 [68.0 to 91.2] | 93.8 [82.8 to 98.7] | 64.4 [48.8 to 78.1] | 95.9 [86.0 to 99.5] | 68.1 [52.9 to 80.9] | 90.2 [78.6 to 96.7] | 47.4 [31.0 to 64.2] | 87.0 [73.7 to 95.1] | 48.5 [39.8 to 57.3] | 70.7 [62.7 to 78.0]

23. Secondary Outcome: Blocking Titers 50 (BT50) of Anti-Norovirus GI.1 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GI.1 VLP antibody titers as measured by HBGA binding assay.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 52 | 51 | 49 | 53 | 45 | 53 | 42 | 52 | 142 | 162
titer | 166.4 [136.0 to 203.6] | 491.4 [397.1 to 608.1] | 135.2 [106.5 to 171.7] | 346.0 [297.5 to 402.3] | 145.0 [108.6 to 193.8] | 531.1 [424.0 to 665.2] | 63.1 [45.3 to 87.9] | 350.1 [273.7 to 447.9] | 202.2 [180.7 to 226.2] | 561.7 [499.2 to 632.1]

24. Secondary Outcome: Blocking Titers 50 (BT50) of Anti-Norovirus GII.4 VLP Antibody Titers (HBGA)
Description: Blocking titers 50 (BT50) of anti-norovirus GII.4 VLP antibody titers as measured by HBGA binding assay.
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 50 | 49 | 46 | 51 | 47 | 54 | 43 | 51 | 136 | 150
titer | 982.1 [652.4 to 1478.4] | 933.6 [678.3 to 1284.9] | 197.1 [119.0 to 326.5] | 514.8 [372.1 to 712.3] | 444.6 [261.9 to 754.8] | 721.8 [510.2 to 1021.1] | 68.5 [44.1 to 106.4] | 282.6 [194.8 to 410.0] | 102.4 [83.1 to 126.1] | 243.9 [203.3 to 292.8]

25. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GI.1 VLP Antibody Titers (HBGA)
Description: as for outcome 18
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 52 | 50 | 49 | 53 | 43 | 50 | 40 | 50 | 137 | 157
ratio | 8.93 [7.58 to 10.53] | 23.07 [18.56 to 28.68] | 7.22 [5.47 to 9.52] | 22.15 [19.06 to 25.73] | 6.10 [4.41 to 8.42] | 24.21 [19.36 to 30.29] | 3.68 [2.64 to 5.13] | 20.01 [15.54 to 25.76] | 11.48 [10.09 to 13.06] | 32.03 [27.38 to 37.47]

26. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of GII.4 VLP Antibody Titers (HBGA)
Description: as for outcome 19
Time Frame: Cohort 1: Day 57; Cohort 2: Day 140
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 49 | 48 | 45 | 49 | 47 | 51 | 38 | 46 | 134 | 147
ratio | 9.31 [6.93 to 12.52] | 12.73 [9.60 to 16.90] | 5.35 [3.94 to 7.28] | 15.95 [12.31 to 20.66] | 8.34 [5.01 to 13.87] | 15.36 [11.26 to 20.96] | 3.91 [2.60 to 5.88] | 17.00 [11.66 to 24.80] | 3.73 [2.84 to 4.90] | 8.13 [6.39 to 10.35]

27. Secondary Outcome: Percentage of Participants With Any Adverse Event (AE) Leading to Withdrawal From the Study
Description: Withdrawal due to an AE will occur if the participant experiences an AE that requires early termination because continued participation imposes an unacceptable risk to the participant's health or the participant is unwilling to continue because of the AE.
Time Frame: Cohort 1: Day 1 up to Day 210; Cohort 2: Day 1 up to Day 293
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
Number analyzed (Participants) | 61 | 59 | 61 | 59 | 60 | 60 | 60 | 60 | 180 | 179
percentage of participants | 0 | 0 | 1.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs 28 days after each vaccination and Serious Adverse Events (SAEs) and AEs leading to trial withdrawal throughout the trial (Up to Day 210 for Cohort 1 and Day 293 for Cohort 2)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1, Group 1: 1 Dose | Cohort 1, Group 1: 2 Doses | Cohort 1, Group 2: 1 Dose | Cohort 1, Group 2: 2 Doses | Cohort 1, Group 2a: 1 Dose | Cohort 1, Group 2a: 2 Doses | Cohort 1, Group 3: 1 Dose | Cohort 1, Group 3: 2 Doses | Cohort 2, Group 4: 2 Doses | Cohort 2, Group 4: 3 Doses
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/61 | 0/59 | 0/60 | 0/60 | 0/60 | 0/60 | 0/180 | 0/179
Serious Adverse Events (participants affected / at risk) | 1/61 | 2/59 | 1/61 | 2/59 | 6/60 | 1/60 | 6/60 | 5/60 | 17/180 | 24/179
Other Adverse Events (participants affected / at risk) | 25/61 | 27/59 | 28/61 | 32/59 | 21/60 | 19/60 | 36/60 | 35/60 | 119/180 | 122/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1: 1 Dose (N=61) | Cohort 1, Group 1: 2 Doses (N=59) | Cohort 1, Group 2: 1 Dose (N=61) | Cohort 1, Group 2: 2 Doses (N=59) | Cohort 1, Group 2a: 1 Dose (N=60) | Cohort 1, Group 2a: 2 Doses (N=60) | Cohort 1, Group 3: 1 Dose (N=60) | Cohort 1, Group 3: 2 Doses (N=60) | Cohort 2, Group 4: 2 Doses (N=180) | Cohort 2, Group 4: 3 Doses (N=179)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 6 | 9
Dengue Fever (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis Media Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular Torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Croup Infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Muscle Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Group 1: 1 Dose (N=61) | Cohort 1, Group 1: 2 Doses (N=59) | Cohort 1, Group 2: 1 Dose (N=61) | Cohort 1, Group 2: 2 Doses (N=59) | Cohort 1, Group 2a: 1 Dose (N=60) | Cohort 1, Group 2a: 2 Doses (N=60) | Cohort 1, Group 3: 1 Dose (N=60) | Cohort 1, Group 3: 2 Doses (N=60) | Cohort 2, Group 4: 2 Doses (N=180) | Cohort 2, Group 4: 3 Doses (N=179)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 15 | 7 | 5 | 8 | 14 | 10 | 23 | 24 | 86 | 92
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4 | 8 | 7 | 0 | 0 | 4 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3 | 3 | 0 | 0 | 5 | 2 | 10 | 15
Pyrexia (General disorders) | 0 | 4 | 4 | 3 | 0 | 0 | 0 | 0 | 6 | 10
Rhinitis (Infections and infestations) | 0 | 0 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 8 | 7
Otitis Media (Infections and infestations) | 0 | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 5 | 2 | 3 | 15 | 11
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 5 | 11 | 11
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 5
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT02153112/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02153112/SAP_001.pdf